CLINICAL TRIAL: NCT03497299
Title: Combining rTMS With Varenicline to Prevent Smoking Lapse in Schizophrenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Yale University (Other); Oregon State University (Other)
Responsible Party: Principal Investigator, Tony George, Chief, Addictions Division, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 003-2017
Record Dates: First submitted 2018-03-29; First posted 2018-04-13 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Tobacco Use Disorder; Schizophrenia; Cognitive Functioning; Craving
Keywords: Schizophrenia; Smoking; Lapse; Varenicline; Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Smoking

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled trial of active versus sham high frequency rTMS to the dorsolateral prefrontal cortex (DLPFC) in patients with schizophrenia who have co-occurring tobacco use disorder. The duration of treatment is 4 weeks and all subjects would receive open label Varenicline 2mg/day. The primary outcome measure is time to lapse to smoking.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigators will have a sham rTMS coil to provide full blinding for the active rTMS condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (20Hz) (Experimental): Active rTMS administered with the MagProX100/R30 stimulator equipped with the B65 active coil for dorsolateral prefrontal cortex (DLPFC) stimulator (MagVenture, Farum, Denmark).The randomization order will be determined by a project scientist from Temerty. While the primary aim of this study is not to treat individuals with tobacco dependence, it is imperative that participants attend weekly study visits in an attempt to achieve end of study (Day 28) tobacco abstinence.
  Interventions: Device: Active rTMS (20Hz)
- Sham rTMS (Sham Comparator): Sham rTMS administered with the MagProX100/R30 stimulator equipped with the B65 placebo coil for DLPFC stimulator (MagVenture, Farum, Denmark). The randomization order will be determined by a project scientist from Temerty. While the primary aim of this study is not to treat individuals with tobacco dependence, it is imperative that participants attend weekly study visits in an attempt to achieve end of study (Day 28) tobacco abstinence.
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS (20Hz) — Repetitive Transcranial Magnetic Stimulation (rTMS) Procedures: On Day 1, participants will be randomly assigned to receive active or sham rTMS using the MagProX100/R30 stimulator equipped with the B65 active/ placebo coil for DLPFC stimulator (MagVenture, Farum, Denmark) for a period of 28 days.
  Arms: Active rTMS (20Hz)
Device: Sham rTMS — Repetitive Transcranial Magnetic Stimulation (rTMS) Procedures: On Day 1, participants will be randomly assigned to receive active or sham rTMS using the MagProX100/R30 stimulator equipped with the B65 active/ placebo coil for DLPFC stimulator (MagVenture, Farum, Denmark) for a period of 28 days.
  Arms: Sham rTMS

SUMMARY:
Tobacco smokers with schizophrenia are known to be resistant smokers, with high rates of smoking and inability to quit in the long-term, often related to smoking relapse. This may relate to problems with frontal lobe function associated with schizophrenia, which make these patients have great difficulty in dealing with smoking withdrawal, urges and cravings. The current study will develop a combination approach that takes advantage of brain stimulation of the frontal lobes (repetitive transcranial magnetic stimulation (rTMS), in combination with the anti-smoking drug varenicline, to prevent smoking lapse using a well-established human laboratory method. Results from this study may have important implications for developing novel treatment approaches for smokers with schizophrenia.

DETAILED DESCRIPTION:
Tobacco smokers with schizophrenia (SWS) represent a subset of smokers with high smoking prevalence compared to the general population, and reduced ability to quit smoking and to resist smoking relapse. There is some evidence that first-line treatments for tobacco use disorder are safe and effective for smoking cessation and smoking relapse-prevention in SWS, but these treatments do not appear to be as effective in smokers with a mental illness as compared to non-psychiatric tobacco smokers. Novel approaches to identify safe and effective treatments using human laboratory models may be an efficient strategy towards this important clinical goal.

The proposed human laboratory study will test the effects of standard pharmacotherapy for tobacco use disorder, the nicotinic partial agonist varenicline, in combination with an established brain stimulation method (repetitive transcranial magnetic stimulation;; rTMS) in SWS. This will allow for the determination of the benefits of combining rTMS with varenciline in SWS using a validated smoking lapse paradigm developed by the collaborator Sherry McKee, Ph.D. at Yale University. The present study represents a novel neuroscience-based strategy for targeting dorsolateral prefrontal cortex (DLPFC) dysfunction in schizophrenia, and is consistent with a target engagement and validation approach as endorsed by NIDA/NIH. Moreover, the subject population the investigators are targeting (SWS) are prone to quit attempt failures and rapid relapse to tobacco smoking, and are in need of novel and effective anti-smoking lapse interventions. The investigators' preliminary data support the use of the combination of varenicline and high-frequency (20 Hz) rTMS to target smoking lapse and craving outcomes in SWS. Accordingly, the investigators believe that the proposed goals, approach and implications for treatment development are substantial and likely to impact positively on clinical treatment research outcomes in this marginalized population of tobacco smokers. Specifically, using a randomized, double-blind, placebo-controlled parallel groups experimental design, the investigators will determine whether the combination of varenicline (2 mg/day) and high-frequency (20 Hz) rTMS versus varenicline and sham rTMS directed to the DLPFC will be superior for the prevention of tobacco smoking lapse behaviors in cigarette smokers with schizophrenia (N=80).

Hypothesis 1 (H1): Active (20 Hz) versus Sham rTMS will increase the time to smoking lapse in combination with varenicline in SWS.

Hypothesis 2 (H2): Active (20 Hz) versus Sham rTMS will improve prefrontal cognition in SWS, and this will be associated with increased ability to resist smoking lapse.

ELIGIBILITY:
Inclusion Criteria:

* smokers with schizophrenia, non-treatment seeking (i.e., not trying to quit as indicated by <7 on the contemplation ladder)
* ages 18-55
* IQ ≥80 on the Weschler Test of Adult Reading
* Fagerstrom Test for Nicotine Dependence (FTND) ≥5
* smoke ≥ 10 cigarettes per day
* must meet SCID for DSM-5 diagnosis criteria for schizophrenia
* must be in stable remission from positive symptoms of psychosis as judged by a PANSS positive score total score <70
* must be receiving a stable dose of antipsychotics for >1month.

Exclusion Criteria:

* substance use (except nicotine or caffeine) in the last month
* a history of alcohol/drug abuse in the 3 months before study enrolment and use of opioids (e.g., meperidine, oxycodone, methadone)
* current use of smoking cessation aids (e.g., nicotine replacement therapy, bupropion or varenicline)
* pregnancy or nursing
* a history of renal insufficiency or a hypersensitivity to varenicline (Chantix®)
* a history of neurological illness like epilepsy or medical condition known to significantly influence neurocognitive function, at the discretion of the PI
* any other medical condition deemed relevant by the PI

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to Smoking Lapse (TTL) | Day 28
  A measure of ability to resist smoking lapse during a 50 minute ad lib cigarette smoking period at Day 28 of the trial in SWS. Higher values indicate increased ability to resist smoking lapse.

SECONDARY OUTCOMES:
Smoking Topography | Day 28 (in comparison to baseline results at Day 0)
  Using the Clinical Research Support System (CReSS), the investigators will assess smoking reinforcement outcomes including total number of puffs smoked per session, total puff volume per cigarette, puffs per cigarette, duration of inter--puff interval, average maximum puff velocity, average puff volume and average puff duration.
Spatial Delayed Response (SDR)/Visuospatial Working Memory (VSWM) Task | Day 28 (in comparison to baseline results at Day 0)
  Subjects focus on a central fixation cross on a computer screen, a dot--shaped cue flashes towards the outer edge of the screen. A delay period then occurs, during which a series of shapes flash in the center of the screen;; the subjects must respond on the spacebar when the diamond shape appears. After the delay, which ranges from 5--30s to assess shorter-- vs. longer--term VSWM, the fixation cross returns and the subject must indicate where they remember seeing the dot. Results are reported as the averaged "distance from target" (cm) for the 16 trials at each delay condition. Duration: 15 minutes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kozak K, Sharif-Razi M, Morozova M, Gaudette EV, Barr MS, Daskalakis ZJ, Blumberger DM, George TP. Effects of short-term, high-frequency repetitive transcranial magnetic stimulation to bilateral dorsolateral prefrontal cortex on smoking behavior and cognition in patients with schizophrenia and non-psychiatric controls. Schizophr Res. 2018 Jul;197:441-443. doi: 10.1016/j.schres.2018.02.015. Epub 2018 Feb 24. PMID 29486960
- [Result] Wing VC, Bacher I, Wu BS, Daskalakis ZJ, George TP. High frequency repetitive transcranial magnetic stimulation reduces tobacco craving in schizophrenia. Schizophr Res. 2012 Aug;139(1-3):264-6. doi: 10.1016/j.schres.2012.03.006. Epub 2012 Mar 29. No abstract available. PMID 22464727